CLINICAL TRIAL: NCT05766501
Title: A Phase 3 Open-label Clinical Study of Doravirine/Islatravir (DOR/ISL [100 mg/0.25 mg]) Once Daily for the Treatment of HIV-1 Infection in Participants Who Previously Received DOR/ISL (100 mg/0.75 mg) QD in a Phase 3 Clinical Study
Brief Title: A Study of Doravirine/Islatravir (DOR/ISL, MK-8591A) for the Treatment of Human Immunodeficiency Virus 1 (HIV-1) Infection in Participants Who Previously Received DOR/ISL (MK-8591A-054)
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 8591A-054; MK-8591A-054 (Other: MSD); 2022-502126-40-00 (Registry Identifier: EU CT); jRCT2051230002 (Registry Identifier: jRCT); U1111-1283-3863 (Registry Identifier: UTN)
Record Dates: First submitted 2023-03-01; First posted 2023-03-13 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: HIV Infection
MeSH Terms: conditions — HIV Infections | interventions — doravirine; islatravir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- DOR/ISL (Experimental): Participants will receive fixed dose combination (FDC) tablet of DOR/ISL (100 mg/0.25 mg) taken once daily (QD) orally from Day 1 to Week 96. After Week 96, eligible participants may continue on DOR/ISL until week 240 or until DOR/ISL becomes commercially accessible, whichever comes first.
  Interventions: Drug: DOR/ISL

INTERVENTIONS:
Drug: DOR/ISL — FDC tablet of 100 mg doravirine (DOR)/0.25 mg islatravir (ISL) taken once daily
  Other Names: MK-8591A; Doravirine/islatravir

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of DOR/ISL in adult participants with HIV-1 who had been previously treated with DOR/ISL in earlier clinical studies. There are no formal hypotheses to be tested in this study.

ELIGIBILITY:
Inclusion Criteria:

* Is currently receiving doravirine/islatravir (DOR/ISL) adult fixed dose combination (FDC) tablet in Merck Sharp & Dohme (MSD)-sponsored clinical studies (MK-8591A-018, -020, and -033 [except for heavily treatment-experienced (HTE) participants]).

Exclusion Criteria:

* Has confirmed HIV-1 RNA ≥200 copies/mL in MSD DOR/ISL (100 mg/0.75 mg) MK-8591A-018 /-020, or at screening for participants entering from DOR/ISL (100 mg/0.75 mg) MK-8591A-033.
* Has confirmatory laboratory findings for cluster of differentiation 4+ (CD4+) T-cell counts or lymphocyte counts in the prior DOR/ISL study that meet criteria for discontinuation of DOR/ISL.
* Is a HTE participant receiving treatment in MK-8591A-019 or -033.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 641 (Actual)
Dates: Start 2023-03-17 (Actual); Primary Completion 2025-10-16 (Actual); Study Completion 2028-09-06 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants with One or More Adverse Event (AE) | Up to 96 Weeks
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study intervention. The percentage of participants who experience an AE through Week 96 will be presented.
Percentage of participants who Discontinue Study Intervention Due to an AE | Up to 96 Weeks
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study intervention. The percentage of participants who discontinue study intervention due to an AE through Week 96 will be presented.

SECONDARY OUTCOMES:
Percentage of Participants with HIV-1 Ribonucleic Acid (RNA) ≥50 copies/mL at Week 96 | Week 96
  The percentage of participants with HIV-1 RNA ≥50 copies/mL at Week 96 will be reported.
Percentage of Participants with HIV-1 RNA <50 copies/mL at Week 96 | Week 96
  The percentage of participants with HIV-1 RNA <50 copies/mL at Week 96 will be reported.
Percentage of Participants with HIV-1 RNA <200 copies/mL at Week 96 | Week 96
  The percentage of participants with HIV-1 RNA <200 copies/mL at Week 96 will be reported
Percentage of Participants with Evidence of Viral Drug Resistance-Associated Substitutions | Up to Week 96
  Viral drug resistance is defined as participants with HIV-1 RNA ≥400 copies/mL and/or genotypic or phenotypic data showing evidence of resistance to the study intervention. The percentage of participants who demonstrate drug resistance through Week 96 will be presented.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (95):
- United States (31):
  - University of Alabama at Birmingham-UAB 1917 Research Clinic ( Site 3104), Birmingham, Alabama
  - Pueblo Family Physicians ( Site 3102), Phoenix, Arizona
  - Pacific Oaks Medical Group ( Site 3123), Beverly Hills, California
  - Kaiser Permanente ( Site 3124), Los Angeles, California
  - Ruane Clinical Research Group, Inc ( Site 3126), Los Angeles, California
  - Mills Clinical Research ( Site 3114), Los Angeles, California
  - University of California Davis Health-Internal Medicine: Infectious Diseases ( Site 3137), Sacramento, California
  - Georgetown University Medical Center ( Site 3130), Washington D.C., District of Columbia
  - Therafirst Medical Center ( Site 3110), Fort Lauderdale, Florida
  - Midway Immunology and Research Center ( Site 3117), Ft. Pierce, Florida
  - AHF The Kinder Medical Group ( Site 3108), Miami, Florida
  - Floridian Clinical Research, LLC ( Site 3133), Miami Lakes, Florida
  - Orlando Immunology Center ( Site 3106), Orlando, Florida
  - Bliss Healthcare Services ( Site 3115), Orlando, Florida
  - CAN Community Health - Sarasota ( Site 3118), Sarasota, Florida
  - Triple O Research Institute, P.A ( Site 3116), West Palm Beach, Florida
  - Augusta University-Infectious Diseases ( Site 3135), Augusta, Georgia
  - Infectious Disease Specialists of Atlanta ( Site 3128), Decatur, Georgia
  - Mercer university, Department of internal medicine-Clinical Research ( Site 3129), Macon, Georgia
  - Chatham County Health Department - Chatham CARE Center-Infectious Disease ( Site 3105), Savannah, Georgia
  - KC CARE Health Center ( Site 3103), Kansas City, Missouri
  - ID Care ( Site 3131), Hillsborough, New Jersey
  - Icahn School of Medicine at Mount Sinai-Clinical and Translational Research Center ( Site 3134), New York, New York
  - Penn Medicine: University of Pennsylvania Health System-Perelman Center for Advanced Medicine ( Site, Philadelphia, Pennsylvania
  - St Hope Foundation ( Site 3121), Bellaire, Texas
  - North Texas Infectious Diseases Consultants, P.A ( Site 3100), Dallas, Texas
  - Texas Centers for Infectious Disease Associates ( Site 3111), Fort Worth, Texas
  - The Crofoot Research Center ( Site 3101), Houston, Texas
  - DCOL Center for Clinical Research ( Site 3119), Longview, Texas
  - Private Practice - Dr. Peter Shalit ( Site 3120), Seattle, Washington
  - Multicare Institute for Research and Innovation ( Site 3127), Spokane, Washington
- Argentina (5):
  - Instituto Oulton ( Site 1004), Córdoba, Córdoba Province
  - Instituto CAICI SRL ( Site 1003), Rosario, Santa Fe Province
  - Helios Salud ( Site 1002), Buenos Aires
  - Fundación Huésped ( Site 1001), Buenos Aires
  - Fundación IDEAA ( Site 1005), Buenos Aires
- Australia (4):
  - Holdsworth House Medical Practice ( Site 1100), Darlinghurst, New South Wales
  - St Vincent's Hospital-IBAC ( Site 1103), Sydney, New South Wales
  - Holdsworth House Medical Practice - Brisbane ( Site 1101), Brisbane, Queensland
  - Prahran Market Clinic ( Site 1102), Melbourne, Victoria
- Canada (6):
  - Hamilton Health Sciences- Urgent Care Centre ( Site 1304), Hamilton, Ontario
  - Maple Leaf Research ( Site 1301), Toronto, Ontario
  - Toronto General Hospital ( Site 1300), Toronto, Ontario
  - Clinique de médecine Urbaine du Quartier Latin ( Site 1305), Montreal, Quebec
  - Clinique Medicale lActuel ( Site 1303), Montreal, Quebec
  - McGill University Health Centre ( Site 1306), Montreal, Quebec
- Chile (6):
  - Clinica Universidad Catolica del Maule ( Site 1405), Talca, Maule Region
  - Biomedica Research Group-Infectology ( Site 1401), Santiago, Region M. de Santiago
  - Pontificia Universidad Catolica de Chile ( Site 1407), Santiago, Region M. de Santiago
  - Universidad de Chile - Hospital Clínico Universidad de Chile-Inmunologia Alergia y VIH ( Site 1400), Santiago, Region M. de Santiago
  - Cardio Sur ( Site 1409), Santiago, Region M. de Santiago
  - Hospital hernan henriquez aravena de temuco-Unidad de Investigación Clínica ( Site 1403), Temuco, Región de la Araucanía
- Colombia (3):
  - Hospital Universitario San Ignacio-Infectious ( Site 1501), Bogotá, Bogota D.C.
  - Clinica Colsanitas S.A, Sede Clínica Universitaria Colombia ( Site 1502), Bogotá, Bogota D.C.
  - Fundación Valle del Lili ( Site 1500), Cali, Valle del Cauca Department
- Israel (4):
  - Rambam Health Care Campus-Institute of Allergy, Clinical Immunology, ( Site 1901), Haifa
  - Hadassah Medical Center-Infecious Disease ( Site 1902), Jerusalem
  - Sheba Medical Center-HIV unit ( Site 1903), Ramat Gan
  - Sourasky Medical Center ( Site 1904), Tel Aviv
- Japan (5):
  - National Hospital Organization Nagoya Medical Center ( Site 2103), Nagoya, Aichi-ken
  - Tokyo Metropolitan Komagome Hospital ( Site 2105), Bunkyo, Tokyo
  - Tokyo Medical University Hospital ( Site 2104), Shinjuku-ku, Tokyo
  - Center Hospital of the National Center for Global Health and Medicine ( Site 2101), Shinjyuku-ku, Tokyo
  - National Hospital Organization - Osaka National Hospital - Institute For Clinical Research ( Site 21, Osaka
- Christchurch Hospital-Infectious Diseases ( Site 2200), Christchurch, Canterbury, New Zealand
- Puerto Rico (2):
  - Clinical Research Puerto Rico ( Site 2400), San Juan
  - HOPE Clinical Research ( Site 2401), San Juan
- Russia (7):
  - Kemerovo Regional Center for the Prevention and Control of AIDS and Infectious Diseases ( Site 2505), Kemerovo, Kemerovo Oblast
  - Krasnoyarsk Regional Center for the Prevention and Control of AIDS ( Site 2504), Krasnoyarsk, Krasnoyarsk Krai
  - Republican Clinical Infectious Hospital ( Site 2500), Saint Petersburg, Leningradskaya Oblast'
  - Moscow Infectious Diseases Clinical Hospital Number 2 ( Site 2506), Moscow, Moscow
  - Scientific Advisory Clinical Diagnostic Center Central Resea-Federal AIDS Center ( Site 2502), Moscow, Moscow
  - Saint-Petersburg Center for Prophylactic of AIDS and Infecti-Saint-Petersburg Center for Prophylact, Saint Petersburg, Sankt-Peterburg
  - Republican Clinical Hospital for Infectious Diseases A.F. Agafonova ( Site 2503), Kazan', Tatarstan, Respublika
- South Africa (9):
  - Josha Research ( Site 2603), Bloemfontein, Free State
  - Perinatal HIV Research Unit (PHRU)-Adult Treatment and Research ( Site 2605), Johannesburg, Gauteng
  - Helen Joseph Hospital-Clinical HIV Research Unit ( Site 2609), Johannesburg, Gauteng
  - Ezintsha-Clinical Research Site ( Site 2607), Johannesburg, Gauteng
  - Private Practice Dr. Marleen de Jager ( Site 2600), Pretoria, Gauteng
  - Wentworth Hospital ( Site 2604), Durban, KwaZulu-Natal
  - Family Clinical Research Unit (Fam-Cru)-Adult Infectious Diseases ( Site 2608), Cape Town, Western Cape
  - Desmond Tutu Health Foundation ( Site 2602), Cape Town, Western Cape
  - Be Part Yoluntu Centre ( Site 2601), Paarl, Western Cape
- Switzerland (6):
  - University Hospital Basel-Infectiology ( Site 2802), Basel, Canton of Basel-City
  - Hôpitaux Universitaires de Genève (HUG)-Infectious Disease Department ( Site 2804), Geneva, Canton of Geneva
  - Cantonal Hospital St.Gallen ( Site 2801), Sankt Gallen, Canton of St. Gallen
  - UniversitätsSpital Zürich ( Site 2800), Zurich, Canton of Zurich
  - Ospedale Regionale di Lugano, Sede Civico-Servizio Malattie Infettive ( Site 2805), Lugano, Canton Ticino
  - Inselspital Bern-Inselspital Infektiologie ( Site 2803), Bern
- Kaohsiung Veterans General Hospital ( Site 2901), Kaohsiung City, Taiwan
- United Kingdom (5):
  - University Hospitals Sussex NHS Foundation Trust ( Site 3004), East Sussex, Brighton And Hove
  - Southmead Hospital ( Site 3003), Bristol, Bristol, City of
  - Royal Free Hospital ( Site 3002), London, England
  - King's College Hospital ( Site 3001), London, London, City of
  - North Manchester General Hospital ( Site 3005), Crumpsall, Manchester

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com/
- See also: Plain Language Summary — https://msd.trialsummaries.com/Study/StudyDetails?id=26164&tenant=MT_MSD_9011